CLINICAL TRIAL: NCT05300867
Title: Robotic Rehabilitation Treatment of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Dr. József Tollár, Head of Neurorehabilitation ,7400 Kaposvár, Tallián Gy. u 20-32, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB2021/10
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Stroke, Acute; Stroke, Ischemic
Keywords: balance; soft exoskeleton; walk; robotic
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Neurological Rehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic (Active Comparator)
  Interventions: Other: Neurorehabilitation
- Controll (Active Comparator)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Neurorehabilitation — Neurorehabilitation with soft exsoskeleton robotic 3-week-long
  Other Names: Rob group
  Arms: Robotic
Other: Physiotherapy — Physiotherapy 3-week-long
  Other Names: Controll groum
  Arms: Controll

SUMMARY:
Storke results in severe deterioration in quality of life and exercise. Severe disorders need to be treated as soon as possible and they need to be rehabilitated quickly in order for motor functions to develop properly. In the acute / subacute phase, patients are given robotic treatment. In addition to the study of mtoros functions, the study of gait and codination is the primary result. Patients treated with soft exoskeleton receive 15 treatments and movement testing is performed continuously. Members of the control group receive standard rehabilitation therapy. After 3 weeks, both groups will participate in a control study and then in a repeat control study at week 6. Our main goal is to compare the results and determine the efficiency of the robotic device.

ELIGIBILITY:
Inclusion Criteria:

post stroke 6MWT : 120> minimum after stroke 3 days

Exclusion Criteria:

Sever heart problem sever demeanor alcoholism drug problems

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Qualiti of life measured by Barthel index | 3 weeks
  quetionnaire
gait/functional test | 3 weeks
  6 minute walk test (m)
gait/functional test | 3 weeks
  10 m walk test (m/s)
balance test | 3 weeks
  Berg balance test
postural control test | 3 weeks
  posturography

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Tollár József, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=robotic+rehabilitation%2C+soft+exoskeleton